CLINICAL TRIAL: NCT06480591
Title: Evaluation of the Pathobiology of CALR-mutated MPN Cells
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Brookdale University Hospital Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00100615; LCI-HEM-MPN-CALR-001 (Other: Atrium Health)
Record Dates: First submitted 2024-06-07; First posted 2024-06-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Thrombosis; JAK2 mutation; CALR mutation
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JAK2 V617F mutation positive MPN patients: Patients with MPN disease with a JAK2 mutation
  Interventions: Other: Blood Draw
- CALR-mutation positive patients: Patients with MPN disease with a CALR mutation
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — The amount of blood that will be collected for this is 50 mL(milliliters), or about 3 ½ tablespoons.

SUMMARY:
The purpose of this study is to understand why there is a greater risk of thrombosis in patients who have the JAK2 mutation as compared to those with CALR mutations.

DETAILED DESCRIPTION:
This biospecimen study is designed to evaluate the expression levels of TLR 2 and TLR 4 on mononuclear cells in CALR mutation positive MPN participants and compare to JAK2 V617F mutation positive MPN patients and healthy controls. Patients who have MPN with the CALR mutation positive will be approached for interest in participating in this study. A research blood collection will occur at any time during the participant's cancer trajectory after enrollment, during a standard of care blood draw. The participant's demographics, MPN subtype, CALR mutation status, history of thrombosis/other medical history, and current, concomitant medications will be collected once. Clinical data will be collected, including results from the CBC with differential, complete metabolic panel (if available), and PT/PTT/INR (if available) drawn closest to the research blood collection. This study will initially open as a single center study at AHWFBCCC.

ELIGIBILITY:
Inclusion Criteria:

* Written (or electronic) informed consent and HIPAA authorization for release of personal health information by participant or his/her legally authorized representative (LAR).
* Age ≥ 18 years at the time of enrollment
* Diagnosis of myeloproliferative neoplasm (MPN) according to 2022 World Health Organization classification of MDS/MPNs
* CALR-positive genetic mutation

Exclusion Criteria:

- Diagnosis of MPN with JAK2 V617F mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in the clinic with MPN with the CALR mutation will be identified and approached for consent.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Expression levels of TLR 2 and TLR 4 | 24 months
  Percentages of mononuclear cells expressing TLR 2 and TLR 4 will be calculated for each participant.

SECONDARY OUTCOMES:
Plasma levels of inflammatory cytokines | 24 months
  Presence and levels of inflammatory cytokines, IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, and TNF-α, will be recorded by multiplex Elisa for each participant.
Plasma levels of inflammatory cytokines following incorporation of TLR ligands | 24 months
  Presence and levels of inflammatory cytokines, IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, and TNF-α, will be calculated for each participant using the in vitro cell culture system.
History of thrombosis | 24 months
  Determined for each participant as a binary variable indicating whether this participant had history of thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Chojecki, MD, Principal Investigator — Atrium Health Levine Cancer
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
Releasing the Individual Participant Data (IPD) is not required to meet the study objectives, and therefore is not planned to be released. Additionally, there is no plan to share data, particularly individual participant data, with anyone who is not already involved in the study